CLINICAL TRIAL: NCT06727539
Title: Prevalence of Hypomineralized Second Primary Molars in a Group of Egyptian Children and Its Association with Molar-Incisor Hypomineralization: a Cross-Sectional Study.
Brief Title: Prevalence of Hypomineralized Second Primary Molars and Its Association with Molar-Incisor Hypomineralization.
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nada Ashraf ElSaeid, Main investigator, Cairo University
Other Study IDs: HSPM in Egyptian children
Record Dates: First submitted 2024-12-09; First posted 2024-12-11 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Molar Incisor Hypomineralisation; Molar Incisor Hypomineralization; Hypomineralization Molar Incisor; Hypomineralization of Enamel
MeSH Terms: conditions — Molar Hypomineralization; Dental Enamel Hypomineralization

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim for thid study is to detect the prevalence of HSPM and the possible association between MIH and HSPM in a group of Egyptian children aged from 6-12 years. The study will also observe the possible etiological factors that might predispose hypomineralization of primary teeth.

To our knowledge, there are no relevant studies that considered the prevalence of HSPM and its possible etiology in Egypt or its association with MIH. So, this study will address this knowledge gap. The possible relationship between HSPM and MIH is highly significant in pediatric dentistry, since the early diagnosis of HSPM as soon as second primary molars erupt makes it possible to initiate more intensive supervision and preventive measures, as these patients are otherwise prone to developing MIH in permanent teeth within a few years.

DETAILED DESCRIPTION:
The highly mineralized tooth enamel consists of nearly 95% of hydroxyapatite crystals and are grouped into highly organized structures called enamel prisms. This structure gives the enamel an exceptional degree of mechanical resistance. Ameloblasts secrete the organic component during tooth formation, after which they polarize and are eliminated from the enamel's surface. Because it no longer contains any living supporting cells, adult enamel is incapable of regeneration.

Enamel formation by ameloblasts passes through several stages: pre-secretory, secretory, transition, maturation, and post-maturation. Depending on whether stage of the ameloblast's life cycle is affected, one can typically find either a normal volume enamel with inadequate mineralization or a fragile and quantitatively deficient enamel. When insufficient mineralization takes place, enamel defects like Molar Incisor Hypomineralization (MIH) and Hypomineralized Second Primary Molar (HPSM) can occur.

MIH is defined as hypomineralization of one to four first permanent molars presenting as well demarcated opacities, qualitative defects of enamel, atypical caries/restorations and extractions due to MIH. It's also frequently associated with the permanent incisors. As of present time, HSPM is defined as hypomineralization of one to four second deciduous molars including the presence of well demarcated opacities, post-eruptive enamel breakdown (PEB), atypical caries or restorations, and extractions due to hypomineralized second primary molars. Recently, these conditions have grabbed the attention of many clinicians across the world mainly because of the worrisome clinical picture and the challenges faced in the management of such conditions.

The etiology of HSPM still remains unclear. Despite that, some potential prenatal, perinatal and postnatal factors have been suggested. Several authors have studied the possible role of risk factors that can cause HSPM based on the medical history given by the parents using structured questionnaires. To date, not a single factor has been found to be an HSPM risk predictor. Furthermore, there is a recall bias potential because all the data obtained from the parents are history-based rather than evaluations of documented medical records.

In addition to this, multiple studies showed a positive correlation between HSPM and MIH, and HSPM being a predictor to MIH. A systematic review and a meta-analysis were done in 2018 aiming to know whether the children with HSPM are likely to have MIH or not and came up with a result that HSPM could be considered as a predictive value to MIH. It was concluded that HSPM can be considered as a specific but not a highly sensitive predictor of MIH which means that the absence of HSPM in primary molars doesn't rule out the potential development of MIH later.

In 2012, a study was done on a group sample of 1,000 Iraqi children ranging between 7-9 years old. A questionnaire-based interview about pregnancy and childhood systemic health history was completed by the mothers. Children with HSPM had greater medical issues, especially in the perinatal stage. The etiology of HSPM is still unknown because no single factor was found to be a likely cause. 94% of children with HSPM have been found to have at least one medical issue, with the likelihood of HSPM increasing with the number of medical issues; 24.5% happening prenatally, 45.3% perinatally, and 9.4% postnatally.

A prospective cohort study was done in 2014 among a 6-year-old group of children to identify possible determinants of HSPM. Data on potential factors that may have occurred during pregnancy and/or the first year of the child's life were gathered using questionnaires and manual, standardized measures (such as weight and length).

A number of pre, peri and postnatal factors have been found to be associated with HSPM.

Those factors included ethnic background, maternal alcohol consumption in pregnancy, low birth weight, and episodes of fever during the first year of the child's life.

In 2014, a study was done on the prevalence and clinical diagnosis of HSPM. Following the diagnostic criteria and the guidelines of the European Academy of Pediatric Dentistry (EAPD), it was concluded that the prevalence of HSPM varied between 4.9 and 9.0 %. HSPM was equally distributed between males and females and between upper and lower arches. It was also concluded that HSPM could be considered as a risk factor and clinical indicator for MIH and no matter how mild the expression of HSPM, it can increase the chance for developing of MIH.

Another study was done on the prevalence and pattern of HSPM among 7 to 10- year-old children in Saudi Arabia. The HSPM prevalence in that study was 5.4% at the child level and 4.8% at the tooth level. Upper right primary second molars were the most affected individual teeth in this study as compared to other primary molars. HSPM cases were found to be more in the maxillary arch as compared to the mandibular arch.

This study also observed there was a positive correlation between HSPM defect extent and increased carious lesion severity.

Concerning the possible association between HSPM and MIH, multiple studies have been done to deeply search into this issue. In 2023, a study was done in South-Western France among 856 children aged between 7-9 years in schools and randomly selected by the Academy of Bordeaux (Ministry of Education). Following the diagnostic criteria for MIH and HSPM of the European Academy of Pediatric Dentistry (EAPD), the risk of having MIH for a child who had HSPM was 52%, while the risk for a child who did not have HSPM was only 15%. The prevalence ratio was 3.4, so the risk of developing MIH was 3.4 times greater if the child had HSPM. In 2023, a cross-sectional study was done on the potential association between MIH and HSPM. The objectives were to evaluate HSPM's predictive value for the MIH and compare the prevalence of HSPM in two child groups; one having MIH and another with no MIH. It also looked into any possible relationships between HSPM severity and MIH severity in a group of children who had both conditions. The prevalence of HSPM in patients who had MIH and who didn't were 37.1% and 11.3%, respectively.

Concerning the relationship between the severity of HSPM and that of MIH in the 79 subjects who had both conditions, mild disease was the most common finding in both MIH and HSPM. 90% of cases of severe HSPM were associated with severe MIH.

A systematic review and meta-analysis were done in 2024 on the possible correlation between HSPM and MIH. Research was conducted in four databases; Embase, PubMed, Web of Science and the Cochrane Library for literature. This meta-analysis included 12 studies with 8,944 children overall. The HSPM group was more likely to experience MIH than the non-HSPM group (OR = 10.90, 95% CI = 4.59-25.89, P <0.05). Every study that was included was of a moderate to high quality.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders will be included
2. Children and adolescents with age group from 6-12 years
3. Participants who agreed to sign rhe informed consent

Exclusion Criteria:

1. Patients having enamel defects like fluorosis, amelogenesis imperfecta and dentinogenesis imperfecta
2. Special health care needs
3. Non-Egyptian children

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study will be done on pediatric patients with the age between 6-12 years old, attending outpatient clinic in the Department of Pediatric Dentistry and Public Health, Cairo university.
Sampling Method: Non-Probability Sample
Enrollment: 825 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Prevalence of HSPM in a group of Egyptian children using EAPD scoring criteria | Baseline
  Prevalence of Hypomineralized Second Primary Molars in a group of Egyptian children using EAPD (European Academy of Pediatric Dentistry) scoring criteria

SECONDARY OUTCOMES:
Correlation of HSPM with MIH | Baseline
  Correlation of Hypomineralized Second Primary Molars with Molar Incisor Hypomineralization using binary outcome (Present/Absent)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marcianes M, Garcia-Camba P, Albaladejo A, Varela Morales M. Predictive Value of Hypomineralization of Second Primary Molars for Molar Incisor Hypomineralization and Other Relationships between Both Developmental Defects of Dental Enamel. J Clin Med. 2023 Aug 25;12(17):5533. doi: 10.3390/jcm12175533. PMID 37685598
- [Background] Estivals J, Fahd C, Baillet J, Rouas P, Manton DJ, Garot E. The prevalence and characteristics of and the association between MIH and HSPM in South-Western France. Int J Paediatr Dent. 2023 May;33(3):298-304. doi: 10.1111/ipd.13040. Epub 2022 Dec 27. PMID 36511101
- [Background] Bekes K, Steffen R, Kramer N. Update of the molar incisor hypomineralization: Wurzburg concept. Eur Arch Paediatr Dent. 2023 Dec;24(6):807-813. doi: 10.1007/s40368-023-00848-5. Epub 2023 Oct 19. PMID 37856065